CLINICAL TRIAL: NCT05082038
Title: Mandibular Full-arch Rehabilitation With Internal Hexagonal and Conical Connection Implants: Randomized Split-mouth Clinical Trial
Brief Title: Mandibular Full-arch Rehabilitation With Internal Hexagonal and Conical Connection Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neodent (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS.I.002
Record Dates: First submitted 2021-09-15; First posted 2021-10-18 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Edentulous Jaw
Keywords: dental implants; oral rehabilitation
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group IF (Other): Two Tapered IF implants will be installed in one side of the mandible
  Interventions: Device: Mandibular partial rehabilitation with IF Tapared implants
- Group CF (Other): Two Tapered IF implants will be installed in the other side of the mandible
  Interventions: Device: Mandibular partial rehabilitation with CF Tapared implants

INTERVENTIONS:
Device: Mandibular partial rehabilitation with IF Tapared implants — 2 IF Tapared Implants (Group IF) on one side of the mandible
  Arms: Group IF
Device: Mandibular partial rehabilitation with CF Tapared implants — 2 CF Tapared Implants (Group CF) on the other side of the mandible
  Arms: Group CF

SUMMARY:
Nuvo Tapered IF (internal hexagonal connection) and CF (conical connextion) Implants were designed for the the oral functional rehabilitation using dental implants, allowing for treatment of patients with different bone qualities.

The aim of the study is to confirm the long-term safety and clinical performance of implants and abutments of Nuvo IF and CF in daily dental practice setting, by means of prospective collection of clinical data in randomized clinical trial using these devices.

Devices will be used , according to manufacturer indications in the IFU. Patients will be followed for 36 months after implant loading.

DETAILED DESCRIPTION:
The study protocol was reviewed and approved by an Ethics Committee (CE) in Brazil. The sample will be prospectively selected and will consist of 18 patients, presenting 18 years of age or more, complete edentulism, who qualify for mandibular rehabilitation by means of full-arch prostheses supported by two Nuvo Tapered IF implants and two Tapered CF implants .Informed consent in writing will be obtained from each patient participating in the study prior to any study related procedure.

Before study site activation, the implants of each patient in the study will be randomly allocated (allocation ratio 1:1), so that each patient receives two implants from each group, on each side of the mandibular arch (Group IF: Tapered Implants with internal hexagonal connection; Group CF: Tapered Implants with conical connection). A blocked randomization list will be generated, where the sequence within block corresponds to the quadrant each group of implants shall be inserted (1:right quadrant; 2: left quadrant). The Randomization List will be kept by the Sponsor in the Trial Master File. Although this study is not blinded, access to the randomization list will not be available to the study centers or to the subjects.

Treatment provided to the subjects will be the responsibility of an appropriately qualified dental practitioners (principal investigator and coinvestigator) to provide the relevant patient care under clinical study conditions, In the mandible, four implants will be placed under local anesthesia and with adequate bone bed preparation, as recommended by the manufacturer, being two Tapered IF implants on one side and two Tapered CF implants on the other, according to the established by the randomization results. The implants will be placed at preferably in an axial position for the medial implants and distally angled for the distal ones, depending on bone availability.

Immediately after implant placement, the final insertion torque shall be recorded. The selection of the prosthetic component and loading protocol (late or immediate) shall be conducted according to the need of each subject and to the manufacturer's instructions (IFU). Thus, implant immediate loading may be performed (at the discretion of the surgeon) when all implants present primary stability of at least 35 N.cm. Maxillary rehabilitation will be performed by means of confection of muco-supported dentures.

Data concerning the studied variables (mandibular rehabilitation) will be collected following the procedures and assessments plan by fulfilling the Case Report Form (CRF), in the following stages: First visit (Screening); TP - Implants placement; T0 - Implant loading; T6, T12, T24 and T36 - 6, 12, 24 and 36 months, respectively, thereafter.

Panoramic radiographs, lateral cephalometric radiographs and computed tomography (CT) scans will be obtained from the region of interest prior to surgery, for the surgical planning. Additionally, standardized digital periapical radiographs will be taken in a usual daily practice frequency, as determined by the investigator: after implants placement (TP - immediately or within 1 week after implant placement) and during the post-operative stages (T0, T6, T12, T24 and T36) to assess the osseointegration process, changes in peri-implant bone level as well as prosthetic settlement and integrity.

ELIGIBILITY:
Inclusion Criteria:

Patients who qualify for mandibular rehabilitation by means of full-arch prostheses supported by two Nuvo Tapered IF implants and two Tapered CF implants

Exclusion Criteria:

Contraindications according to the Instructions for Use of the device will be applied, as follows:

* Signs of allergy or hypersensitivity to the chemical ingredients of the material: titanium;
* Presence of acute inflammatory or infectious processes in live tissue;
* Unsuitable bone volume and/or quality;
* Systemic complications or diseases such as: bone metabolism disorders, blood clotting disorders, unsuitable healing capacity, insufficient oral hygiene, incomplete jawbone growth, patient uncooperative and not motivated, abuse of drugs or alcohol, psychosis, prolonged functional disorders which resist any treatment with medications, xerostomia, weakened immunological system, diseases which require the use of steroids, endocrinological diseases, pregnancy.

The research does not involve minors, or women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Periimplant bone level change | up to 36 months
  Amount of Periimplant bone level change 36 months after loading.

SECONDARY OUTCOMES:
Implant survival rate | up to 36 months
  Survival will be defined as no loss of the implant at each follow-up
Prosthetic survival | 6, 12, 24 and 36 months
  Prosthetic survival will be assessed as the final prosthesis remaining in situ at each follow-up.
Soft tissue evaluation | up to 36 months
  visible plaque index, maginal bleeding index, bleeding on probing, gingival index, keratinized tissue height measurements
Patient satisfaction | up to 36 months
  The Portuguese translation of OHIP-EDENT questionnaire will be used to assess Oral Health Related Quality of Life (OHRQoL), as a measure of patient satisfaction with treatment.
Clinician satisfaction | up to 36 months
  The assessment will be performed by means of a questionnaire using a visual analog scale (VAS) in the form of a 10 cm horizontal line, where 0 (left end) indicates minimum satisfaction and 10 (right end) indicates maximum satisfaction
Adverse events | up to 36 months
  Determined by inquiring with the patient and clinical evaluation
Device deficiences | up to 36 months
  Determined by inquiring with the patient and clinical evaluation
Implant success rate | up to 36 months
  * Absence of persisting subjective discomfort such as pain, foreign body perception and or dysaesthesia (painful sensation);
  * Absence of a recurrent periimplant infection with suppuration (infection is termed recurrent if observed at two or more follow-up visits after the treatment with systemic antibiotics);
  * Absence of implant mobility on manual palpation;
  * Absence of any continuous periimplant radiolucency.
Prosthetic success rate | up to 36 months
  Success will be defined as the prosthesis that remained unchanged and did not require any intervention

CONTACTS AND LOCATIONS:
Overall Officials: Waleska Caldas, PhD, Study Chair — Neodent
Locations (1):
- Mattias Sartori Consultoria Em Odontologia, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No